CLINICAL TRIAL: NCT01718808
Title: Cetuximab Monotherapy and Cetuximab Plus Capecitabine as First-line Treatment in Elderly Patients With KRAS- and BRAF Wild-type Metastatic Colorectal Cancer. A Multicenter Phase II Trial
Brief Title: Cetuximab for Elderly Patients With mCRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FU for 3 years from randomization as initially planned is stopped as we do not expect any changes to the endpoints in the future after one year of FU.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/10
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; KRAS; BRAF; Wild-type Metastatic; Cetuximab; Capecitabine; Phase II Trial; Elderly Patients
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Cetuximab (Active Comparator): Cetuximab 500 mg/m2 every 2 weeks
  Interventions: Drug: Cetuximab
- Arm B: Cetuximab and Capecitabine (Active Comparator): Cetuximab 500 mg/m2 every 2 weeks plus Capecitabine 1000 mg/m2 (*) bid d1-14 every 3 weeks
  * 750 mg/m2 if creatinine-clearance 30-50 ml/min
  Interventions: Drug: Cetuximab; Drug: Capecitabine

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 500 mg/m2 every second week (days 1, 15, 29, etc.) until progression or unacceptable toxicity
  Other Names: Erbitux
Drug: Capecitabine — Capecitabine 1000 mg/m2 bid p.o. (750 mg/m2 if creatinine clearance 30-50 ml/min according to Cockroft-Gault formula, on days 1-14 every 3 weeks, restart on day 22
  Other Names: Xeloda
  Arms: Arm B: Cetuximab and Capecitabine

SUMMARY:
OBJECTIVE: The objective of the trial is to judge on the benefit obtained by an upfront cetuximab treatment delivered as monotherapy or as part of a combination treatment with capecitabine in vulnerable elderly patients selected for V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) wild-type and B-type Raf kinase (BRAF) wild-type metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Primary endpoint: If in a treatment arm the number of patients alive and without progression at 12 weeks is 17 or more, this arm will be considered promising, otherwise not promising. Additionally, a two-sided 95% confidence interval for the difference in Progression free survival (PFS) rates between the two arms will be calculated.

Secondary endpoints and patient characteristics:

* Laboratory values may be expressed as the absolute values (continuous variables) or/and as grading (ordinal categorical variables).
* Generally for each categorical variable the results will be summarized by frequencies and percentages. For response rates 95% Clopper-Pearson confidence intervals will be calculated.
* For each adverse event, the results will be summarized by frequencies and percentages of different grades among all cycles as well as by frequencies and percentages of the within-patient worst grades
* For each continuous variable the results will be summarized by descriptive statistics.
* Time-to-event variables will be presented by Kaplan-Meier curves and summarized by medians and 95% confidence intervals.
* All analysis will be done by treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before any trial specific treatment
* Histological proven diagnosis of colorectal cancer, metastatic or inoperable advanced, not amenable to curative therapy
* Measurable disease, defined as at least one lesion (outside of irradiated areas) that can be measured in at least one dimension as ≥ 10 mm (≥ 15 mm in case of lymph nodes) according to RECIST v1.1
* Tumour with wild-type KRAS and wild-type BRAF gene
* No previous systemic chemotherapy for metastatic disease (previous adjuvant chemotherapy is allowed if completed >6 months before randomization, previous rectal radio-chemo therapy if completed >1 month before randomization)
* WHO performance status 0 or 1
* Age >75 years; or: age ≥ 70 years with at least one of the following factors:
* Any functional dependence as measured by Instrumental Activities of Daily Life (IADL). Significant comorbidity according to the Cumulative Illness Rating Scale for geriatric patients (CIRS-G; any severe comorbidity > grade 3 or a total score > 5 qualifies)
* Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Bilirubin ≤ 2.0 x Upper Limit of Normal (ULN) (unless known Gilbert-Meulengracht syndrome), aspartate aminotransferase (AST)<2.5xULN
* Calculated creatinine clearance ≥ 30 ml/min. (according to the formula of Cockcroft-Gault)
* Patient is able to swallow oral medication
* Baseline Quality of Life forms have been completed

Exclusion Criteria:

* Documented or suspected cerebral and/or leptomeningeal metastases (no cerebral baseline imaging required in asymptomatic patients)
* Risk of rapid deterioration due to tumor symptoms or tumor complications
* Synchronous or prior malignancy other than adequately treated non-melanomatous skin cancer or in situ carcinoma of the cervix, other malignancies unless disease free > 2 years
* Prior anti-EGFR (Epidermal Growth Factor Receptor) antibody therapy
* Severe or uncontrolled cardiovascular disease (e.g. acute coronary syndromes, cardiac failure NYHA (New York Heart Association) III or IV, clinically relevant myopathy, history of myocardial infarction within the last 12 months, significant arrhythmias)
* Concurrent severe uncontrolled medical illness (judged by the investigator) which could impair the ability of the patient to participate in the trial (e.g. uncontrolled infection, uncontrolled diabetes mellitus, active autoimmune disease)
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drug
* Definite contraindications for the use of corticosteroids or antihistamines as premedication
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome or history of inflammatory intestinal disease, or other disease which could alter drug absorption
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out QL forms, or interfering with compliance with oral drug intake
* Any concomitant drugs contraindicated for use with the trial drugs according to the Swissmedic approved product information
* Concurrent treatment with other experimental drugs or other anti-cancer therapy and/or treatment in a clinical trial within 30 days prior to randomization

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival in week 12 | in week 12
  A progression event is defined as (whichever occurs first):
  * Progressive disease (PD) assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
  * Death of any cause
  * Starting of second line treatment
  * No tumor assessment 85 days (+/- 7 days) after registration which shows stabilisation or response Patients without tumor assessment at week 12 but with a later assessment showing absence of progression without subsequent treatment will be counted as a progression free at week 12

SECONDARY OUTCOMES:
Quality of life (QL) | Baseline, in week 7, 13 and 19
Adverse events (CTCAE v 4.0) | Adverse events are assessed by Common terminology criteria for adverse events (CTCAE) v4.0. From randomization until 30 days after end of treatment (estimated up to 2 years).
Overall Response (OR) | Before start of treatment. In week 13 and every 12 weeks up to 2 years.
Progression free survival (PFS) | PFS will be calculated sustained from randomization until documented PD or death, whichever occurs first (estimated up to 2 years).
Overall Survival (OS) | Overall survival will be calculated from randomization until death (estimated up to 2 years).
Overall treatment utility (OTU) (predefined composite endpoint including clinical benefit, tolerability and acceptability of the treatment) | Until week 19.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Kienle, MD, Study Chair — Kantonsspital Graubünden; Roger von Moos, MD, Study Chair — Kantonsspital Graubünden; Ralph Winterhalder, MD, Study Chair — Luzerner Kantonsspital; Dieter Köberle, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (14):
- Switzerland (14):
  - Universitaetsspital-Basel, Basel
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Hopital Fribourgeois, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Muensterlingen, Muensterlingen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - Klinik Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No